CLINICAL TRIAL: NCT04007133
Title: Evaluation of Statin Compliance of Patients With Non-insulin-dependent Diabetes
Brief Title: Statin Compliance of Patients With Non-insulin-dependent Diabetes
Acronym: DIOS
Status: Terminated | Type: Observational
Why Stopped: The study was conducted in the context of a medical thesis with a deadline.
Sponsor: Lille Catholic University (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0064
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Non-insulin-dependent Diabetes
Keywords: Non-insulin-dependent diabetes; Statins; Compliance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients: Patients with non-insulin-dependent diabetes, taking statins for at least 1 month
  Interventions: Other: Girerd test

INTERVENTIONS:
Other: Girerd test — This is a simple and quick questionnaire, composed of 6 questions with a binary yes/no answer. It allows to assess the degree of compliance with the prescribed treatment to better identify the constraints related to the treatment.

SUMMARY:
The diabetic population has an increased cardiovascular risk compared to the general population.

Hydroxymethylglutaryl-CoA reductase (HMG-CoA reductase) inhibitors, or "statins", are considered as the standard treatment for hypercholesterolemia.

Many patients with non-insulin-dependent diabetes are prescribed with statins, both for primary prevention, before the first cardiovascular event, and as secondary prevention, to avoid recurrence.

However, compliance to these drugs may be difficult due to polypharmacy, side effects (myalgia) or tiredness.

The purpose of this study is to determine the compliance of diabetic patients with statins searching for important factors which could favor adherence.

DETAILED DESCRIPTION:
The diabetic population has an increased cardiovascular risk compared to the general population. The mortality of people with diabetes due to ischemic heart disease is multiplied by 2.2, and when is due to cerebrovascular disease by 1.8 compared to those patients without diabetes. Hydroxymethylglutaryl-CoA reductase (HMG-CoA reductase) inhibitors, or "statins", are considered as the standard treatment for hypercholesterolemia.

Statins have been shown to be effective in reducing the risk of cardiovascular events, each 1 mmol decrease in LDL cholesterol reduces the risk of cardiovascular events by 21% at 5 years.

Many patients with non-insulin-dependent diabetes are prescribed with statins, both for primary prevention, before the first cardiovascular event, and for secondary prevention, to avoid recurrence.

However, compliance with these drugs may be difficult due to polypharmacy, side effects (myalgia) or tiredness. Indeed, the persistence of statin use, one year after its prescription, is estimated at 70% in the general population. However, there are no data in the French population, and in particular on French diabetic patients for whom the cardiovascular risk is increased compared to the general population.

The purpose of this study is to determine the compliance of diabetic patients with statins searching for important factors which could favor adherence.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* With non-insulin-dependent diabetes, taking statins for at least 1 month (to assess compliance)
* Hospitalized in the Diabetology Day Hospital of the Saint Philibert Hospital
* In capacity to answer the Girerd test
* Patient who has been informed and not opposed to the study

Exclusion Criteria:

* Patient's refusal to participate in the study
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with non-insulin-dependent diabetes, taking statins for at least 1 month
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Compliance rate with statin measured by the Girerd test | Day 0
  This is a simple and quick questionnaire, composed of 6 questions with a binary yes/no answer. It allows to assess the degree of compliance with the prescribed treatment and thus to better identify the constraints related to the treatment. The score varies from 0 to 6 depending on the presence of "yes". 0 "yes": Good compliance, more than 3 "yes": non compliance.

SECONDARY OUTCOMES:
Compliance rate with statin according to the type of prevention | Day 0
  Type of prevention (primary/secondary) and compliance rate measured by the Girerd test
Compliance rate with statin according to risk factors | Day 0
  Link between compliance rate measured by Girerd test and potential factors analyzed: age, sex, polypharmacy, duration of diabetes, no previous cardiovascular history, no prior dyslipidemia, blood LDL level, duration of statin intake, modalities of treatment preparation, understanding of the benefits of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Lille Catholic Hospitals, Lomme, Nord, France

IPD SHARING:
Plan to Share IPD: No